CLINICAL TRIAL: NCT05424445
Title: Orally Administered Misoprostol Solution (Cytotec®) Versus Orally Administered Misoprostol as a Tablet (Angusta®) for Induction of Labor in Women With Mixed Parity and an Unfavorable Cervix, a Randomized Controlled Trial.
Brief Title: MISOBEST - Orally Misoprostol Solution (Cytotec®) Versus Orally Misoprostol as a Tablet (Angusta®) for Induction of Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tove Wallström, MD, PhD, senior consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2020-000663-23
Record Dates: First submitted 2022-01-21; First posted 2022-06-21 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Induced Vaginal Delivery
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Masking Description: Due to the nature of the study, comparing the same drug but in different preparations, blinding is not deemed feasible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytotec® (Experimental): IOL with misoprostol oral solution (Cytotec®) 25 ug every second hour, up to eight doses, or until painful contractions are obtained. Thereafter IOL will proceed according to clinical practice.
  Interventions: Drug: Misoprostol
- Angusta® (Active Comparator): IOL with misoprostol oral tablets (Angusta®) 25 ug every second hour, up to eight doses, or until painful contractions are obtained. Thereafter IOL will proceed according to clinical practice.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Women presenting at the study site with an indication for IOL will receive written and oral information about the study. They will have the opportunity to ask questions. If the woman agrees to participate and is deemed eligible, she will sign informed consent. The Swedish national guidelines regarding the method of IOL will be followed. Women will have an abdominal palpation to exclude malpresentation, a CTG, and a digital cervical exam to establish bishop score (BS) prior to inclusion (as per clinical practice). Randomization will be performed by the attending physician, midwife or study coordinator. Randomization will be by opening numbered opaque sealed envelopes in sequential order containing the randomization code. There are no restrictions for use of other medications. All concomitant medication will be recorded in the CRF.

SUMMARY:
The aim of the study is to evaluate efficacy of the cervical ripening of misoprostol administration in oral tablet, Angusta® compared with the off-label solution of misoprostol (Cytotec®) for induction of labor (IOL). Since there is a large cost difference between the preparations (Angusta® is 43 times more expensive than Cytotec®) it is, from a socio-economic perspective, of great interest to evaluate if Angusta can be replaced by Cytotec.

DETAILED DESCRIPTION:
In Sweden as in most other countries, the rate of induction of labor (IOL) has steadily increased, peaking at 27% of all deliveries in 2020. Due to recently published studies showing decreased perinatal mortality with IOL at 41 instead of 42 gestational weeks, national guidelines have changed to offering all pregnant women reaching 41 weeks IOL, which will increase induction rates and subsequent cost of IOL for medication further.

Spontaneous onset of labor is usually preferred, as it generally means lower risk of complications compared to IOL. If delivery needs to be induced in women with an unfavorable cervical status, an oral solution of misoprostol is a safe and inexpensive method that is easy to control and provides a high success rate of vaginal deliveries with a very low risk of hyper stimulation. Since the preparation of misoprostol (Cytotec®) has been used off-label with the solution being prepared locally at every unit, the profession has been looking for alternatives. Angusta® 25 ug tablets is the alternative that has been developed and approved but without being compared to the oral solution of misoprostol, the most commonly used method for IOL in Sweden. In addition, Angusta® is 43 times more expensive (1011 SEK compared to 23.60 SEK for Cytotec® for eight doses) considering "a typical induction" for primiparous women. Both methods are currently in use in clinical practice in Sweden.

A recent study conducted in Sweden 2020 shows that the Area Under the Curve (AUC) for the concentration in the blood of misoprostol after administration of 25 ug Cytotec® po compared to Angusta® 25ug po differs . The AUC is 32.9% higher with Cytotec® compared to Angusta®. The lower AUC for Angusta® may result in lower efficacy and time to delivery. However, this is unknown. The reason for this difference may be that a greater proportion of misoprostol is absorbed buccally and/or sublingually with use of misoprostol as a solution compared to when it is used as a tablet. Misoprostol has significantly different effect on uterine contractility depending on method of administration(1). Thus, using Angusta® may result in negative health economic outcomes due to higher price and in addition, a longer time spent in the delivery unit. No comparison of these two formulations has been performed in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestations
* Cephalic presentation
* ≥37-42+0 weeks of gestation
* Unfavorable cervix score BS <6 in nulliparous women and <5 in parous women
* All participating women in the studies will receive oral and written information and must give informed consent before participation

Exclusion Criteria:

1. Inability to understand the study information written in Swedish or English
2. Previous hysterotomy (scar in the uterine myometrium)
3. Non-reassuring cardiotocography (CTG) on admission (the door-test, first 20 minutes of registration of CTG).
4. Hypersensitivity to the active substance
5. If active labor has started
6. When oxytocin infusion is already used
7. Placenta previa
8. Renal failure (GFR <15 ml/min/1.73 m2).
9. Any condition or circumstance due to which the investigator considers it is not in the best interest of subject to participate in the study or the inclusion of a subject risks negatively impacting the scientific or ethical integrity of the clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 884 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery within 24 hours (VD 24) rate as difference in proportions in each group according to intention-to-treat (ITT), and per protocol. | Time point for extraction of data: immediately after the intervention/procedure/surgery
  VD24 - (yes/no) is a dichotomous variable extracted from medical records.

SECONDARY OUTCOMES:
Proportion of vaginal deliveries (VD) in total. | Time point for extraction of data: immediately after the intervention/procedure/surgery.
  VD (dichotomous, electronic patient records).
The induction-to-vaginal delivery time. | Time point for extraction of data:immediately after the intervention/procedure/surgery.
  Induction-to-delivery interval (continuous, electronic patient records).
The mean number of doses of each preparation. | Time point for extraction of data: immediately after the intervention/procedure/surgery.
  Number of doses of each preparation (electronic patient records).
The proportion of neonates with Apgar <7 at 5 minutes. | Time point for extraction of data: immediately after the intervention/procedure/surgery.
  Children with Apgar <7 at 5 minutes (electronic patient records).
Postpartum bleeding (PPH) >1000 ml. | Time point for extraction of data: immediately after the intervention/procedure/surgery.
  PPH >1000 ml (electronic patient records.
The proportion of women with hyper stimulation defined as painful contractions. exceeding 5 in 10 minutes with CTG abnormalities. | Time point for extraction of data: immediately after the intervention/procedure/surgery.
  Cardiotocography electronic patient records.
Cost-effectiveness. | Time point for extraction of data: immediately after the intervention/procedure/surgery.
  Cost effectiveness calculated as ICER (incremental cost effectiveness ratio). The ICER considers changes in effectiveness as well as cost of treatment and was established using the formula: [Cost of Intervention-Cost of Standard treatment]/ [Effectiveness Intervention-Effectiveness of Standard treatment]. The intervention is Cytotec® and the control is Angusta®.
  The parameters included in the calculation are: Normal birth (no complications), normal birth( with complications), assisted delivery, Cesarean section ( no complications), Cesarean section (with complications, misoprostol as a tablet ((Angusta®) and as a solution (Cytotec®),oxytocin infusion, Midwife - hospital appointment (unit cost/minute), Consultant (unit cost/minute), Cost of perinatal death, Hospital admission for induction (hospital hotel costs), Cost of admission to neonatal nursery (per day) according to a study (8), in the book chapter in NICE guidelines, induction of labor.

CONTACTS AND LOCATIONS:
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stephansson O, Petersson K, Bjork C, Conner P, Wikstrom AK. The Swedish Pregnancy Register - for quality of care improvement and research. Acta Obstet Gynecol Scand. 2018 Apr;97(4):466-476. doi: 10.1111/aogs.13266. Epub 2017 Dec 14. PMID 29172245
- [Background] Wennerholm UB, Saltvedt S, Wessberg A, Alkmark M, Bergh C, Wendel SB, Fadl H, Jonsson M, Ladfors L, Sengpiel V, Wesstrom J, Wennergren G, Wikstrom AK, Elden H, Stephansson O, Hagberg H. Induction of labour at 41 weeks versus expectant management and induction of labour at 42 weeks (SWEdish Post-term Induction Study, SWEPIS): multicentre, open label, randomised, superiority trial. BMJ. 2019 Nov 20;367:l6131. doi: 10.1136/bmj.l6131. PMID 31748223
- [Background] Tang J, Kapp N, Dragoman M, de Souza JP. WHO recommendations for misoprostol use for obstetric and gynecologic indications. Int J Gynaecol Obstet. 2013 May;121(2):186-9. doi: 10.1016/j.ijgo.2012.12.009. Epub 2013 Feb 19. PMID 23433680
- [Background] Amini M, Reis M, Wide-Swensson D. A Relative Bioavailability Study of Two Misoprostol Formulations Following a Single Oral or Sublingual Administration. Front Pharmacol. 2020 Feb 12;11:50. doi: 10.3389/fphar.2020.00050. eCollection 2020. PMID 32116725
- [Derived] Svensk E, Bessfelt E, Brismar Wendel S, Kopp Kallner H, Wallstrom T. Misoprostol as Oral Solution or Oral Tablet for Induction of Labour (MISOBEST): A Randomised Controlled Non-Inferiority Trial. BJOG. 2025 Feb;132(3):288-296. doi: 10.1111/1471-0528.17986. Epub 2024 Oct 23. PMID 39440409